CLINICAL TRIAL: NCT01535053
Title: A Phase III Randomized Trial of Pulse Actinomycin-D Versus Multi-day Methotrexate for the Treatment of Low-Risk Gestational Trophoblastic Neoplasia
Brief Title: Dactinomycin or Methotrexate in Treating Patients With Low-Risk Gestational Trophoblastic Neoplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GOG Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0275; NCI-2012-00250 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000725211; PGOG-0275_A08PAMDREVW01; GOG-0275; GOG-0275 (Other: NRG Oncology); GOG-0275 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Choriocarcinoma; FIGO Stage I Gestational Trophoblastic Tumor; FIGO Stage II Gestational Trophoblastic Tumor; FIGO Stage III Gestational Trophoblastic Tumor; Hydatidiform Mole
MeSH Terms: conditions — Choriocarcinoma; Hydatidiform Mole | interventions — Dactinomycin; Leucovorin; Methotrexate; merphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (dactinomcin) (Experimental): Patients receive dactinomycin IV over 15 minutes on day 1.
  Interventions: Biological: Dactinomycin; Other: Quality-of-Life Assessment
- Arm II (leucovorin calcium and methotrexate) (Active Comparator): Patients receive methotrexate IM on days 1, 3, 5, and 7 and leucovorin calcium PO on days 2, 4, 6, and 8 OR single agent methotrexate IV on days 1-5.
  Interventions: Drug: Leucovorin Calcium; Drug: Methotrexate; Other: Quality-of-Life Assessment

INTERVENTIONS:
Biological: Dactinomycin — Given IV
  Other Names: Actinomycin A IV; Actinomycin C1; Actinomycin D; Actinomycin I1; Actinomycin IV; Actinomycin X 1; Actinomycin-[thr-val-pro-sar-meval]; Cosmegen; DACT; Dactinomycine; Lyovac Cosmegen; Meractinomycin
  Arms: Arm I (dactinomcin)
Drug: Leucovorin Calcium — Given PO
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Arm II (leucovorin calcium and methotrexate)
Drug: Methotrexate — Given IV and IM
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Arm II (leucovorin calcium and methotrexate)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized phase III trial studies how well methotrexate works compared to dactinomycin in treating patients with low-risk gestational trophoblastic neoplasia. Drugs used in chemotherapy, such as methotrexate and dactinomycin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether methotrexate is more effective than dactinomycin in treating gestational trophoblastic disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the hypothesis that treatment with multi-day methotrexate is inferior to treatment with pulse actinomycin-D (dactinomycin) in patients with low-risk gestational trophoblastic disease with respect to complete response.

SECONDARY OBJECTIVES:

I. To describe the frequency of post protocol surgical treatment for each arm. II. To describe the frequency of post protocol multi-agent chemotherapy treatment for each arm.

III. To compare multi-day methotrexate to actinomycin-D with respect to frequency and severity of adverse events in patients with low-risk gestational trophoblastic neoplasia.

IV. To investigate the impact of treatment on overall quality-of-life (QOL) and explore the influence of treatment on issues such as body image, sexual functioning, and patient-reported side effects and disruption.

V. To assess whether uterine artery pulsatility index (UAPI) can provide independent prognostic information predictive of single-drug resistance.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive dactinomycin intravenously (IV) over 15 minutes on day 1.

ARM II: Patients receive methotrexate intramuscularly (IM) on days 1, 3, 5, and 7 and leucovorin calcium orally (PO) on days 2, 4, 6, and 8 OR single agent methotrexate IV on days 1-5.

In both arms, treatment repeats every 14 days for up to 20 courses* in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for 1 year and then every 3 months for 1 year.

NOTE: * Patients will be treated for three courses after human chorionic gonadotropin (hCG) < 5 mIU/mL or until evidence of treatment failure (biologic progression), disease progression, or unacceptable toxicity despite dose modifications. Upon normalization of hCG (< 5 mIU/mL), patients will be treated with three additional courses.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet International Federation of Gynecology and Obstetrics (FIGO) stage I, II, or III criteria for low-risk gestational trophoblastic neoplasia (GTN): post molar GTN or choriocarcinoma (as defined below); patients may have had a second curettage but must still meet GTN criteria below:

  * Post molar GTN

    * For the purposes of this study, patients must have undergone evacuation of a complete or partial hydatidiform mole and then meet the criteria for GTN defined as:

      * A < 10% decrease in the hCG level using as a reference the first value in the series of 4 values taken over a period of 3 weeks (> 50 mIU/ml minimum) OR
      * A > 20% sustained rise in the hCG taking as a reference the first value in the series of 3 values taken over a period of 2 weeks (> 50 mIU/ml minimum) OR
      * A persistently elevated hCG level a period of 6 months or more following the initial curettage (> 50 mIU/ml minimum)
  * Choriocarcinoma

    * Histologically proven non-metastatic choriocarcinoma OR
    * Histologically proven metastatic choriocarcinoma if the metastatic site(s) is restricted to one (or more) of the following: vagina, parametrium, or lung
* World Health Organization (WHO) risk score 0-6
* Patients must be willing to practice effective contraception for the duration of the study
* White blood cell count (WBC) >= 3,000 cells/mcL
* Granulocytes >= 1,500/mcL
* Platelets >= 100,000/mcL
* Creatinine =< 2.0 mg/dcL
* Bilirubin =< 1.5 x institutional normal
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x institutional normal
* Alkaline phosphatase =< 3 x institutional normal
* Patients who have met the pre-entry requirements
* Before enrolling a patient, the institution must verify the availability of an adequate supply of methotrexate for a full course of therapy
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients who do not have GTN
* Patients with non-gestational choriocarcinoma
* Patients who have previously been treated with cytotoxic chemotherapy; however, patients who received prior low-dose methotrexate for treatment of an ectopic pregnancy will be eligible for this study
* Patients who have received prior pelvic radiation
* Patients with placental-site trophoblastic tumor (PSTT) or epithelioid trophoblastic tumor (ETT)
* Patients with Gynecologic Oncology Group (GOG) performance status of 3 or 4
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients whose circumstances at the time of study entry do not permit completion of the study or required follow-up
* Patients who wish to breast-feed during treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-06-18 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian C Schink, Principal Investigator — NRG Oncology
Locations (289):
- United States (267):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Low Country Cancer Care, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Cancer Care Partners LLC, Mishawaka, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Monongalia Hospital, Morgantown, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (2):
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
- Japan (11):
  - Tohoku University School of Medicine, Sendai, Aoba-ku
  - Kure National Hospital, Kure, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - University of the Ryukyus Hospital-Col Health Scnc, Nakagami-gun, Okinawa
  - Hiroshima University Hospital, Hiroshima
  - Kindai University, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - Tottori University, Tottori
- South Korea (8):
  - Samsung Medical Center, Seoul, Korea
  - Catholic University of Korea-Seoul Saint Mary's Hospital, Seoul, Korea
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Gachon University Gil Hospital, Incheon
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul
- Weston Park Hospital, Sheffield, England, United Kingdom

REFERENCES:
- [Derived] Schink JC, Filiaci V, Huang HQ, Tidy J, Winter M, Carter J, Anderson N, Moxley K, Yabuno A, Taylor SE, Kushnir C, Horowitz N, Miller DS. An international randomized phase III trial of pulse actinomycin-D versus multi-day methotrexate for the treatment of low risk gestational trophoblastic neoplasia; NRG/GOG 275. Gynecol Oncol. 2020 Aug;158(2):354-360. doi: 10.1016/j.ygyno.2020.05.013. Epub 2020 May 24. PMID 32460997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 6/18/2012and closed to accrual prematurely on 9/20/2016 by the sponsor due to slow accrual.
Pre-assignment Details: Sites declared in advance which of 2 methotrexate regimens they would follow for patients who received a random treatment allocation to the methotrexate arm. Randomization is stratified by country (US, Canada, Japan, Korea, Australia, United Kingdom, etc.) and Multi-day methotrexate regimen (8- or 5-day) used by the participating site.
Groups:
- Regimen I (Dactinomycin): IV pulse actinomycin-D (1.25mg/m2 ) every 14 days. (2mg max dose)
- Regimen II (Methotrexate): institutional preference of either:
  * IV methotrexate (0.4 mg/kg) daily for 5 days every 14 days. (25mg max daily dose) OR
  * IM methotrexate (50mg) on Days 1, 3, 5, 7 (4 doses per cycle) with Leucovorin (15mg) on Days 2, 4, 6, 8. Repeat every 14 days.
Period: Overall Study
Arm/Group | Regimen I (Dactinomycin) | Regimen II (Methotrexate)
Started | 29 | 28
Completed | 28 (treated for 3 cycles after hCG <5mIU/ml or until biologic,disease progression, unacceptable toxicity) | 26 (treated for 3 cycles after hCG <5mIU/ml or until biologic,disease progression, unacceptable toxicity)
Not Completed | 1 | 2
Not completed — Ineligible | 1 | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen I (Dactinomycin) | Regimen II (Methotrexate) | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Customized [Count of Participants; unit: Participants]
  10-19 years | 1 | 1 | 2
  20-29 years | 14 | 11 | 25
  30-39 years | 11 | 11 | 22
  40-49 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 24 | 50
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 16 | 19 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response
Description: Complete Response is defined as 3 consecutive bi-weekly values of hCG<5 over a minimum of 4 weeks of normal hCG values with no values greater than 5 mIU/ml
Time Frame: hCG testing is performed prior to each cycle to treatment until treatment is completed, up to 10 months. For patients who have responded to treatment hCG must be obtained every 4 weeks for 1 year after completing treatment.
Population: Eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Regimen I (Dactinomycin) | Regimen II (Methotrexate)
Number analyzed (Participants) | 28 | 26
percentage of participants | 78.6 [59.0 to 91.7] | 88.5 [69.8 to 97.6]

2. Secondary Outcome: Number of Participants With CTCAE v4 Graded Adverse Events With Low-risk Gestational Trophoblastic Neoplasia by Arm
Description: Maximum grade of physician assessed adverse events reported during treatment
Time Frame: Assessed throughout the treatment period and within 2-4 weeks after discontinuation of treatment
Population: Eligible and treated patients
Measure: Number; unit: participants
Arm/Group | Regimen I (Dactinomycin) | Regimen II (Methotrexate)
Number analyzed (Participants) | 28 | 26
participants
  Grade 1 | 7 | 4
  Grade 2 | 14 | 10
  Grade 3 | 6 | 10
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

3. Secondary Outcome: The Number of Participants With Post Protocol Surgical Treatment for Each Arm.
Time Frame: Anytime during post treatment follow-up for up to 2 years from study entry.
Population: Non-responding eligible patients in follow-up
Measure: Number; unit: participants
Arm/Group | Regimen I (Dactinomycin) | Regimen II (Methotrexate)
Number analyzed (Participants) | 7 | 5
participants | 0 | 0

4. Secondary Outcome: The Number of Participants With Post Protocol Multi-agent Chemotherapy Treatment for Each Arm.
Time Frame: Anytime during post treatment follow-up for up to 2 years from study entry.
Population: Non-responding eligible patients in follow-up
Measure: Number; unit: participants
Arm/Group | Regimen I (Dactinomycin) | Regimen II (Methotrexate)
Number analyzed (Participants) | 7 | 5
participants | 0 | 0

5. Secondary Outcome: Patient-reported Quality of Life (QOL) at Baseline
Description: Patient reported quality of life was measured with the Functional Assessment of Cancer Therapy - Generic (FACT-G). The FACT-G is a scale for assessing general QOL of cancer patients. It consists of four subscales: Physical Well Being, Functional Well Being, Social/Family Well-Being, and Emotional Well-Being. Each item in the FACT-G was scored using a 5-point scale (0=not at all; 1=a little bit; 2=somewhat; 3=quite a bit; 4=very much). For the negative statements, reversal was performed prior to score calculation. According to the FACIT measurement system, a subscale score was the summation of the individual item scores if more than 50% of subscale items were answered. When unanswered items existed, a subscale score was prorated by multiplying the mean of the answered item scores by the number of items in the subscale. The FACT-G score is calculated as the sum of the subscale scores. The FACT-G score ranges 0-108. A larger score suggests better QOL.
Time Frame: Prior to cycle 1
Population: Provided baseline QOL questionnaire
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Regimen I (Dactinomycin) | Regimen II (Methotrexate)
Number analyzed (Participants) | 27 | 27
units on a scale | 82.3 (2.7) | 81.9 (3.3)

6. Secondary Outcome: Patient-reported Quality of Life (QOL) After Baseline Visit.
Description: as for outcome 5
Time Frame: Prior to cycle 3 (4 weeks after cycle 1 if off study treatment prior to cycle 3). Prior to cycle 5, Prior to cycle 7, 26 weeks after starting study treatment.
Population: Provided baseline and ≥1 follow-up assessments
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Regimen I (Dactinomycin) | Regimen II (Methotrexate)
Number analyzed (Participants) | 27 | 27
units on a scale
  Pre-cycle 3 | 78.3 (2.3) | 81.6 (2.7)
  Pre-cycle 5 | 75.5 (3.3) | 78.9 (2.8)
  Pre-cycle 7 | 85.0 (2.7) | 84.5 (2.2)
  26 weeks | 91.2 (2.9) | 90.9 (2.9)

ADVERSE EVENTS:
Time Frame: Through Study Treatment and up to 30 days after discontinuing treatment.
Description: Participants listed in the all-cause mortality include all enrolled. Participants in the Serious Adverse Event and Other Adverse Events include all eligible AND treated. Therefore, the number of participants listed in the all-cause mortality is larger than the serious adverse event and other adverse event tables.
Arm/Group | Regimen I (Dactinomycin) | Regimen II (Methotrexate)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/26
Other Adverse Events (participants affected / at risk) | 27/28 | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen I (Dactinomycin) (N=28) | Regimen II (Methotrexate) (N=26)
Appendicitis (Infections and infestations) | 0 | 1
Psychiatric Disorders - Other (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen I (Dactinomycin) (N=28) | Regimen II (Methotrexate) (N=26)
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 1
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1 | 3
Anemia (Blood and lymphatic system disorders) | 13 | 15
Palpitations (Cardiac disorders) | 1 | 1
Cardiac Disorders - Other (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 4
Hearing Impaired (Ear and labyrinth disorders) | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 2 | 0
Eye Disorders - Other (Eye disorders) | 0 | 3
Watering Eyes (Eye disorders) | 0 | 4
Eye Pain (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 0 | 1
Blurred Vision (Eye disorders) | 4 | 3
Dry Eye (Eye disorders) | 0 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 12 | 11
Diarrhea (Gastrointestinal disorders) | 7 | 7
Vomiting (Gastrointestinal disorders) | 8 | 6
Stomach Pain (Gastrointestinal disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 10 | 6
Oral Dysesthesia (Gastrointestinal disorders) | 1 | 0
Mucositis Oral (Gastrointestinal disorders) | 12 | 20
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 0 | 1
Gingival Pain (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 20 | 16
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 1
General Disorders And Administration Site Conditio (General disorders) | 3 | 0
Pain (General disorders) | 0 | 2
Malaise (General disorders) | 3 | 1
Localized Edema (General disorders) | 0 | 1
Flu Like Symptoms (General disorders) | 1 | 2
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Edema Limbs (General disorders) | 1 | 0
Edema Face (General disorders) | 0 | 1
Fatigue (General disorders) | 18 | 15
Fever (General disorders) | 2 | 1
Chills (General disorders) | 1 | 1
Allergic Reaction (Immune system disorders) | 0 | 1
Infections And Infestations - Other (Infections and infestations) | 4 | 1
Upper Respiratory Infection (Infections and infestations) | 0 | 1
Vulval Infection (Infections and infestations) | 0 | 1
Skin Infection (Infections and infestations) | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 1
Vaginal Infection (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Investigations - Other (Investigations) | 1 | 0
Weight Gain (Investigations) | 0 | 2
Platelet Count Decreased (Investigations) | 3 | 4
Hemoglobin Increased (Investigations) | 1 | 0
Ggt Increased (Investigations) | 1 | 1
Neutrophil Count Decreased (Investigations) | 5 | 7
White Blood Cell Decreased (Investigations) | 4 | 6
Aspartate Aminotransferase Increased (Investigations) | 2 | 1
Alkaline Phosphatase Increased (Investigations) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 7
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal And Connective Tissue Disorder - O (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 8 | 5
Facial Muscle Weakness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Psychiatric Disorders - Other (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Personality Change (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 6
Depression (Psychiatric disorders) | 1 | 1
Confusion (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 2
Urinary Retention (Renal and urinary disorders) | 1 | 0
Urinary Tract Pain (Renal and urinary disorders) | 1 | 0
Urinary Frequency (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 3
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 1 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 6 | 7
Vaginal Dryness (Reproductive system and breast disorders) | 0 | 1
Perineal Pain (Reproductive system and breast disorders) | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 2 | 0
Irregular Menstruation (Reproductive system and breast disorders) | 1 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 5 | 3
Vaginal Inflammation (Reproductive system and breast disorders) | 0 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 5
Thromboembolic Event (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hot Flashes (Vascular disorders) | 3 | 1
Flushing (Vascular disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Early closure leading to non-compliance and small numbers of subjects analyzed. Study cannot be considered terminated because some participants are still being examined for follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT01535053/Prot_SAP_000.pdf